CLINICAL TRIAL: NCT02354521
Title: NUTRITION SUPPORT DURING PEDIATRIC CRITICAL ILLNESS - 2ND MULTICENTER, INTERNATIONAL COHORT STUDY OF BARRIERS AND OUTCOMES
Brief Title: Nutrition Support During Pediatric Critical Illness - 2nd Multicenter, International Cohort Study
Acronym: PINS2
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Nilesh M. Mehta, Associate Professor of Anesthesia, Critical Care, Boston Children's Hospital
Other Study IDs: X-10 11 0569
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Nutrition
Keywords: Protein; Mechanical ventilation; Children; Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: NO INTERVENTIONS

SUMMARY:
An observational, point-prevalence cohort study of nutrition therapies in critically ill children in PICUs across the world. Baseline information will be collected including PICU and hospital demographics and characteristics (e.g. age, diagnostic category, PRISM score, weight, height) of critically ill children requiring mechanical ventilation in the PICU. Nutrition practices such as route of nutrition, kilocalorie and protein levels prescribed and received, interruptions, etc., will be collected on a daily basis from PICU admission onwards, for a maximum of 10 days. Data on clinical outcomes (e.g. duration of mechanical ventilation, PICU stay, hospital stay, acquired infections) will be collected up to 60 days after admission to the PICU. The main objective of the study is to examine the association between energy and protein intake adequacy (in relation to the prescribed goals for these nutrients) and 60-day mortality in mechanically ventilated children.

DETAILED DESCRIPTION:
Nutrition Support can prevent complications associated with malnutrition and when used appropriately has a positive influence on clinically important outcomes, such as length of stay, morbidity and mortality. Making decisions regarding the most effective and safe nutrition support can be challenging, and consequently considerable variation exists in nutrition support practices in PICUs.

This is a multicenter prospective cohort study of nutritional practices in mechanically ventilated children from a representative sample of medium to large (at least 8 ICU beds) PICUs in North America and participating centers across other countries. The investigators will invite centers in all 9 US Census regions, at least 3 Canadian Provinces and PICUs with 8 or more beds from across the world. Participating sites will be recruited through the PALISI network (of more than 66 PICUs), by disseminating study information through national nutrition (e.g. ASPEN) and critical care societies (e.g. (SCCM), and e-mailing individual healthcare providers.

Patient selection criteria: All children (ages 1month to 18 years) admitted to the PICU, who require mechanical ventilatory support with anticipated duration of stay longer than 48 hours will be eligible for data collection. Data collection for each eligible patient will be continued for a total of 10 days or until discharge from the PICU (if earlier) until a minimum of 15 patients (maximum 40 patients) are accrued per site. The investigators anticipate recruitment of 500 patients.

The trained dietitians (or a designated research nurse) at participating centers will use a validated web-based remote data capture tool to record details of nutritional intake. An instruction package describing data collection methods in detail will be provided. Following a training period, beginning on the 'going live' date, the dietitian or designated coordinator at participating centers will simultaneously enter relevant data online using a secure website.

Nutritional variables including the energy and protein goals prescribed by the local nutrition team, actual daily macronutrient delivery achieved, route of delivery, frequency and duration of feeding interruptions, and use of adjunctive drugs, will be recorded. Prescribed protein goals for each subject will be compared to the recommended daily protein in the 2005 DRI and the 2009 A.S.P.E.N. age-based guidelines. The end point for nutritional data collection is 10 days or discharge from the PICU, whichever was sooner. The energy and protein intake adequacy will be calculated as the percentage of the prescribed goal that was actually delivered and an average adequacy over the PICU stay up to 10 days was derived.

The primary outcome for this study is 60-day patient mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 month to 18 yrs
* PICU anticipated stay longer than 48 hours, on mechanical ventilatory support

Exclusion Criteria:

* Patients who were not ventilated within the first 48 hours of admission to PICU
* On compassionate care toward end-of-life
* Those enrolled in any other nutritional intervention trial will be excluded

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (age 1 month to 18 yrs) admitted to the PICU with anticipated stay longer than 48 hours, and who require mechanical ventilatory support.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
60-day mortality | 60 days

SECONDARY OUTCOMES:
Acquired infections | PICU stay
  Acquired infections include ventilator associated pneumonia, urinary tract infection and catheter associated blood stream infection during the PICU stay.
Ventilator free days | 28 days

REFERENCES:
- [Background] Mehta NM, Bechard LJ, Cahill N, Wang M, Day A, Duggan CP, Heyland DK. Nutritional practices and their relationship to clinical outcomes in critically ill children--an international multicenter cohort study*. Crit Care Med. 2012 Jul;40(7):2204-11. doi: 10.1097/CCM.0b013e31824e18a8. PMID 22564954
- [Derived] Mehta NM, Bechard LJ, Zurakowski D, Duggan CP, Heyland DK. Adequate enteral protein intake is inversely associated with 60-d mortality in critically ill children: a multicenter, prospective, cohort study. Am J Clin Nutr. 2015 Jul;102(1):199-206. doi: 10.3945/ajcn.114.104893. Epub 2015 May 13. PMID 25971721